CLINICAL TRIAL: NCT02427893
Title: An Exploratory Study of the Immunological Effects of Vemurafenib and Cobimetinib, Administered Alone and in Combination, in Subjects With Advanced BRAF V600E/K Mutant Melanoma
Brief Title: Trial of Vemurafenib and Cobimetinib in Patients With Advanced BRAFV600 Mutant Melanoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no patients were enrolled
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1517; IRB00051085 (Other: JHMIRB)
Record Dates: First submitted 2015-03-27; First posted 2015-04-28 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
Keywords: immunotherapy; Vemurafenib; Cobimetinib
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Ten patients begin Vemurafenib monotherapy, after 10 days, begin combination therapy by adding Cobimetinib.
  Interventions: Drug: Cobimetinib; Drug: Vemurafenib
- Cohort 2 (Active Comparator): Ten patients begin Cobimetinib monotherapy, after 10 days, begin combination therapy by adding Vemurafenib.
  Interventions: Drug: Cobimetinib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — A potent and highly selective inhibitor of MEK1 and MEK2, central components of the RAS/RAF pathway.
  Other Names: GDC-0973, XL518
Drug: Vemurafenib — A low molecular weight, orally available inhibitor of the activated form of the BRAF serine-threonine kinase enzyme, which is commonly found in melanoma
  Other Names: RO5185426, PLX4032, or RG7204

SUMMARY:
This trial explores the immunologic effects of vemurafenib (BRAF inhibitor) and cobimetinib (MEK inhibitor), administered alone and in combination, to patients with advanced BRAF V600E/K mutant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Signed HIV testing consent
* Life expectancy ≥ 12 weeks
* Able to swallow pills
* ECOG performance status 2 or less
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function
* Negative urine pregnancy test within 7 days prior to commencement of dosing in premenopausal women
* Histological diagnosis of unresectable AJCC stage III or stage IV, BRAFV600E/K mutant melanoma
* Measurable disease
* Accessible tumor that can be biopsied
* Naive to targeted therapy (Prior immune-based therapy in the adjuvant setting or for advanced disease will be allowed if >2 weeks from study entry)

Exclusion Criteria:

* Active systemic infection
* Active autoimmune disease or history of known or suspected autoimmune disease
* Active brain metastases or leptomeningeal metastases
* Treatment with any immunomodulatory medication within 4 weeks of initiation of study therapy.
* Positive test for hepatitis B virus
* Positive test for hepatitis C virus
* Positive test for human immunodeficiency virus (HIV)
* Pregnant, lactating or breast feeding women
* Localized radiation therapy within the last 14 days
* History of malabsorption
* No consumption of the following within 7 days prior to start of treatment:

  * St. John's wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer)
  * Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor
* History or evidence of cardiovascular risk
* History or evidence of retinal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of cobimetinib monotherapy and combination vemurafenib/cobimetinib in subjects with advanced melanoma. | 2 years
  compare immunologic changes described above with the development of study treatment-related adverse events. For example, severity or extent of rash from cobimetinib (a well-described dermatologic toxicity of MEK inhibitors) may be compared to levels of intratumoral immune activation assessed by one or more of the parameters.

SECONDARY OUTCOMES:
Anti-tumor activity of cobimetinib monotherapy and combination vemurafenib/cobimetinib in subjects with advanced melanoma. | 2 years
  compare immunologic changes described above with therapeutic outcomes, including CR, PR, SD, and PD measured by RECIST 1.1. For example, tumor regression may be correlated with levels of intratumoral immune activation or expression of immune checkpoints assessed by one or more of the parameters

CONTACTS AND LOCATIONS:
Overall Officials: Evan J Lipson, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States